CLINICAL TRIAL: NCT00983736
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of Two Doses of Tramadol Hydrochloride Orally Disintegrating Tablets in Male Subjects With Premature Ejaculation
Brief Title: Study to Evaluate Efficacy and Safety in Male Subjects With Premature Ejaculation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated because of recruitment difficulties.
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BVF-324-302
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2010-11

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Tramadol Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol Hydrochloride — 89 mg or a lesser dose of 62 mg if side effects are experienced one tablet at least two hours before sexual intercourse (maximum of one tablet every 20 hours).
  Subject will take the study drug for about 27 weeks.
  Arms: Active
Drug: Placebo — 89 mg or a lesser dose of 62 mg if side effects are experienced one tablet at least two hours before sexual intercourse (maximum of one tablet every 20 hours).
  Subject will take the study drug for about 27 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to test an experimental drug therapy called Tramadol Hydrochloride (HCl) Orally Disintegrating Tablets (ODT) ("Tramadol HCl ODT" or the "study drug"). The patient and the patient's partner are being asked to be in this clinical trial because they have a condition called Premature Ejaculation.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for study participation if all of the following criteria are met:

1. Male subject and female partner to provide written informed consent prior to the performance of any study-specific procedures;
2. Candidates will be male subjects aged 18-65 years inclusive, with lifelong premature ejaculation ("lifelong" is defined as starting at the time the subject became sexually active) with an IELT of ≤120 seconds as documented at Visit 2.
3. History of premature or rapid ejaculation, determined by following criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM IV TR):

   1. Persistent or recurrent ejaculation with minimal sexual stimulation before, on, or shortly after vaginal insertion and before the person wishes it, taking into account factors that affect duration of the excitement phase such as age, novelty of the sexual partner or situation and recent frequency of sexual activity
   2. The disturbance causes marked distress or interpersonal difficulty
   3. The premature ejaculation is not due exclusively to the direct effects of a substance (ab)use
4. In a stable, monogamous, heterosexual relationship (> 6 months).
5. Willing and able to take study medication as directed at least 2 hours prior to sexual intercourse according to protocol;
6. Subject willing and able to complete the therapeutic trial, all sexual behavior logs, IELT assessments, questionnaires and interviews:
7. Female sexual partner willing and able to complete the therapeutic trial, all sexual behavior logs, IELT assessments, questionnaires and interviews;
8. Able to understand the study procedures, complete the assessments, and communicate with study personnel;
9. Subject and partner willing and able to engage in vaginal intercourse at least three times between visits to yield at least three events of vaginal intercourse ;
10. Subject and partner willing to use a reliable contraceptive method during the trial period if the partner is not menopausal;
11. Partner willing to take pregnancy tests at Visits 1 and 2
12. Subject willing to list and document prescription and non-prescription drug use during the study;
13. Have a negative urine drug screen at Visits 1 and 2;
14. Be in good general health as determined by medical history and physical examination and expected by the Investigator to complete the study as designed.

Exclusion Criteria:

Subjects are not eligible for study participation if any of the following criteria are met:

1. Premature ejaculation attributable to situational or relationship issues;
2. Evidence or a history of other significant psychiatric disorder as defined as requiring therapy or medication;
3. Subjects who in the Investigator's opinion are at significant risk of suicide.
4. Physical illnesses

   i.History of seizures

   ii.Prostatitis (current)

   iii.Urethritis or other urinary tract infections (current)

   iv.Prior genital surgery (other than vasectomy or circumcision)

   v.Uncontrolled Diabetes mellitus

   vi.Respiratory Depression

   vii.Thyroid disease

   viii.Chronic moderate to severe neurological disease

   ix.Significant heart disease treated with cardiac drugs

   x.Chronic liver disease

   xi.Chronic kidney disease

   xii.History of cardiovascular disease (myocardial infarction, congestive heart failure, angina, coronary artery disease or stroke)

   xiii.Known to be a carrier of the hepatitis B surface antigen, hepatitis C virus antibody, and/or immunodeficiency virus-1 and/ or 2 antibodies

   xiv.Other disorder that may cause sexual dysfunction
5. Other sexual dysfunction:

   i.Erectile dysfunction. As defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV TR), the diagnostic criteria for male erectile disorder (302,72) erectile dysfunction includes:

   A.Persistent or recurrent inability to attain, or to maintain until completion of the sexual activity, an adequate erection.

   B.The disturbance causes marked distress or interpersonal difficulty. ii.Primary reduced sexual desire unrelated to premature ejaculation
6. Sexual intercourse usually less than once per week;
7. Partner sexual dysfunction (for example dyspareunia or other conditions considered relevant);
8. Current use of dapoxetine;
9. Current use of any tramadol;
10. Sensitivity to phenylketone;
11. Any history of abuse of prescription opioids and/or illicit/illegal addictive drugs;
12. Has a known hypersensitivity to heparin or history of heparin induced thrombocytopenia;
13. Use of medication, within the preceding 30 days, with potential to cause sexual dysfunction: (See Appendix 2 for a list of excluded medications)

    i.Antidepressants - all types

    ii.Antipsychotic medication

    iii.Antihypertensive medication, unless on a stable dose > 6 months

    iv.Hormonal drugs

    v.Chemotherapy

    vi.Others: cimetidine, clofibrate,quinidine
14. Recent psychotropic drug use (within the past 30 days);
15. A history of alcohol abuse or dependence within the past 6 months as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV TR);
16. Initiation of psychosexual counseling during the screening, baseline or treatment periods;
17. Partner positive pregnancy test at Visit 1 or 2;
18. History of clinically significant intolerance or a known hypersensitivity to tramadol, such that treatment with it is contraindicated;
19. The Investigator anticipates that the subject will be unable to comply with the protocol;
20. Received any investigational drug within 30 days prior to Visit 1 or is scheduled to receive an investigational drug during the course of this study;
21. Has preplanned surgery or procedures that would interfere with the course of the study.
22. A family member (other than the female partner), a staff member, or relative of a staff member..
23. Significant laboratory abnormality as determined by the Investigator at Visit 1;
24. Significant ECG abnormality at Visit 1 as determined by the Investigator;
25. Any other illnesses, conditions or practices that in the Investigator's opinion could interfere with the collection and/or interpretation of study results (couples using the "Withdrawal Method" of birth control will be excluded from the study).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Increase in IELT (Intravaginal ejaculatory time) | Per attempt at sexual intercourse

SECONDARY OUTCOMES:
Efficacy of using Tramadol for Premature Ejaculation | At each attempt

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nyiradi, MD, Principal Investigator — Mediroyal Prevention Center
Locations (48):
- Bulgaria (10):
  - MHAT, Urology Clinic, 8A G. Kochev Str., Pleven
  - MHAT Plovdiv, Plovdiv
  - MHAT Sveti Georgl Plovdiv, Urology Clinic, 66 Peshtersko Shosse Str., Plovdiv
  - MHAT Ruse, Urology Depart., 2 Nezavisimost Str., Rousse
  - CCB SAI Ministry of Interior, 79A, Skobelev Blvd., Sofia
  - MHAT Aleksandrovska, Urology Clinic, 1st, Georgi Sofiski Str., Sofia
  - MHAT Doverie, Urology Depart, 2 Ovcha Kupel, Quadrant 18, Sofia
  - SHAT Endocrinology "Academic Ivan Penchev", Sofia
  - MHAT "Sveta Anna" Varna Urology Clinic, Varna
  - MHAT DR Stefan Cherkezov, Veliko Tarnovo
- Czechia (9):
  - Urazova Nemocnice v Brne, Brno
  - Andrologicka Ambulance, Hradec Králové
  - Psychiatricke Oddeienf and Sexuologicka Ambulance, Pardubice
  - Soukroma Sexuologicka a Psychiatricka Ambulance, Pilsen
  - Androgeos S. R. O., Prague
  - Fakultni Thomayerova Nemocnice, Prague
  - TH Klinika S.R.O., Prague
  - Urologicka Klinika S.R.O., Prague
  - Medicentrum Olomouc, S.T.O., Řepčín
- Hungary (8):
  - Allami Egeszegugyi Kozpont (State Health Center), Budapest
  - Donatella 99BT Private Healthcare Center, Budapest
  - Erector Clinic Uro-Szexologiai Centrum, Budapest
  - Semmelwiis Egyetem Urolgiai Klinika, Budapest
  - Mediroyal Prevention Center, Györe
  - Soproni Erzesebet Oktato Korhaz, Györe
  - Szegeci Tudomanyegyetem Altalanos Orvostudomanyl Kar Urologial Kinika, Kálvária
  - Sandor Egeszegogyl Kozpont, Vinár
- Poland (12):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Klinika Urologii Uniwersytet Medyczny, Gdansk
  - Nzoz Vip-Med, Gdynia
  - Indywidualna Specjalistyczna Praktyka Lekarska, Katowice
  - Prywatna Praktyka Seksuologiczna, Lodz
  - Indywidualna Specjalistyczna Praktyka Lekarska, Poznan
  - Indywidualna Specjalistyczna Praktyka Lekarska Polozniczo-Ginekologiczno-Seksuologiczna, Szczecin
  - Nzoz 'Constans-Med', Todz
  - MEDEA Specialistyczny, Warsaw
  - Poradnia Seksuologii i Patologll Wiezl Miedzyludzkich, Warsaw
  - Szaleckl Lempicki Spolka Partnersaka Lekarzy Urologow, Warsaw
  - Gabinet Lekanski Dr. Med. Ryszard Smolinski, Wroclaw
- Romania (9):
  - Spitalul Clinic de Urgenta "Sf. Loan", Urologie, Bucharest
  - Spitalul Clinic de Urgenta Militar Central "Dr. Carol Davila", Bucharest
  - Spitalul Clinicl Prof. Theodor Burghele, Sectia Urologie II, Bucharest
  - Uro-andro-Med SRL, Bucharest
  - Provita 2000 SRL, Constanța
  - Spitalul Clinic Judetean de Urgenta Craiova, Sectia Urologie, Craiova
  - Spitalul Clinic Constantin Bucuras, Judetul Timis
  - Spitalul Clinic Judetean de Urgenta Oradea, Urologie, Oradea
  - Centrul Medical 'SF. Pantelimon', Cabinetul de Urologie, Pantelimon

REFERENCES:
- [Derived] Bar-Or D, Salottolo KM, Orlando A, Winkler JV; Tramadol ODT Study Group. A randomized double-blind, placebo-controlled multicenter study to evaluate the efficacy and safety of two doses of the tramadol orally disintegrating tablet for the treatment of premature ejaculation within less than 2 minutes. Eur Urol. 2012 Apr;61(4):736-43. doi: 10.1016/j.eururo.2011.08.039. Epub 2011 Aug 30. PMID 21889833